CLINICAL TRIAL: NCT02579382
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Multi-center Study to Evaluate the Safety and Efficacy of GS-9620 in Combination With Tenofovir Disoproxil Fumarate (TDF) for the Treatment of Subjects With Chronic Hepatitis B and Who Are Currently Not on Treatment
Brief Title: Study to Evaluate the Safety, Tolerability, and Efficacy of Vesatolimod in Combination With Tenofovir Disoproxil Fumarate (TDF) in Adults With Chronic Hepatitis B (CHB) Infection Who Are Currently Not Being Treated
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-283-1062; 2015-002017-30 (EudraCT Number)
Record Dates: First submitted 2015-10-15; First posted 2015-10-19 (Estimated); Results first posted 2020-05-18 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Chronic Hepatitis B
Keywords: HBV; Hepatitis; Liver Disease
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis; Liver Diseases | interventions — Tenofovir; vesatolimod

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- TDF + placebo (Placebo Comparator): Main Study Phase: Tenofovir disoproxil fumarate (TDF) 300 mg tablets orally once daily for up to 48 weeks + placebo administered orally once a week (every 7 days) for 12 doses.
  Optional Treatment Extension Phase: At Week 48 participants had the option to continue TDF 300 mg tablets orally once daily up to Week 144.
  Interventions: Drug: TDF; Drug: Placebo
- TDF + Vesatolimod 1 mg (Experimental): Main Study Phase:TDF 300 mg tablets orally once daily for up to 48 weeks + vesatolimod 1 mg tablet orally once a week (every 7 days) for 12 doses.
  Optional Treatment Extension Phase: At Week 48 participants had the option to continue TDF 300 mg tablets orally once daily up to Week 144.
  Interventions: Drug: TDF; Drug: Vesatolimod
- TDF + Vesatolimod 2 mg (Experimental): Main Study Phase: TDF 300 mg tablets orally once daily for up to 48 weeks + vesatolimod 2 mg tablet orally once a week (every 7 days) for 12 doses.
  Optional Treatment Extension Phase: At Week 48 participants had the option to continue TDF 300 mg tablets orally once daily up to Week 144.
  Interventions: Drug: TDF; Drug: Vesatolimod
- TDF + Vesatolimod 4 mg (Experimental): Main Study Phase: TDF 300 mg tablets orally once daily for up to 48 weeks + vesatolimod 4 mg tablet orally once a week (every 7 days) for 12 doses.
  Optional Treatment Extension Phase: At Week 48 participants had the option to continue TDF 300 mg tablets orally once daily up to Week 144.
  Interventions: Drug: TDF; Drug: Vesatolimod

INTERVENTIONS:
Drug: TDF — 300 mg tablets administered orally once daily
  Other Names: Viread®
Drug: Vesatolimod — Tablets administered orally once a week (every 7 days) for 12 doses
  Other Names: GS-9620
  Arms: TDF + Vesatolimod 1 mg; TDF + Vesatolimod 2 mg; TDF + Vesatolimod 4 mg
Drug: Placebo — Placebo administered orally once a week (every 7 days) for 12 doses
  Arms: TDF + placebo

SUMMARY:
The primary objectives of this study are to evaluate the safety, tolerability, and efficacy of vesatolimod (formerly GS-9620) in adults with chronic hepatitis B (CHB) infection who are currently not being treated.

ELIGIBILITY:
Key Inclusion Criteria:

* Adult males or females between the ages of 18-65
* Chronic hepatitis B virus (HBV) infection
* HBV deoxyribonucleic acid (DNA ) ≥ 2000 IU/mL at screening

Key Exclusion Criteria:

* Extensive bridging fibrosis or cirrhosis
* Received oral antiviral treatment for HBV or prolonged therapy with immune-modulators or biologics within 3 months of screening
* Co-infection with hepatitis C virus (HCV), human immunodeficiency virus (HIV) or hepatitis D virus (HDV)
* Chronic liver disease other than HBV
* Lactating or pregnant females or those that wish to become pregnant during the course of the study

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2015-11-10 (Actual); Primary Completion 2017-01-16 (Actual); Study Completion 2019-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (21):
- United States (9):
  - Los Angeles, California
  - Palo Alto, California
  - San Diego, California
  - San Francisco, California
  - Honolulu, Hawaii
  - Catonsville, Maryland
  - Boston, Massachusetts
  - Flushing, New York
  - Philadelphia, Pennsylvania
- Toronto, Ontario, Canada
- Kowloon, Hong Kong
- Italy (4):
  - Bologna
  - Milan
  - Pisa
  - San Giovanni Rotondo
- Grafton, Auckland, New Zealand
- South Korea (2):
  - Daegu
  - Seoul
- Taiwan (2):
  - Dalin
  - Kaohsiung City
- London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Agarwal K, Ahn SH, Elkhashab M, Lau AH, Gaggar A, Bulusu A, Tian X, Cathcart AL, Woo J, Subramanian GM, Andreone P, Kim HJ, Chuang WL, Nguyen MH. Safety and efficacy of vesatolimod (GS-9620) in patients with chronic hepatitis B who are not currently on antiviral treatment. J Viral Hepat. 2018 Nov;25(11):1331-1340. doi: 10.1111/jvh.12942. Epub 2018 Aug 22. PMID 29851204
- [Result] Younossi ZM, Stepanova M, Janssen H, Agarwal K, Nguyen MH, Gane EJ, et al. The impact of treatment of chronic hepatitis B (CHB) on patient reported outcomes (PROs). Poster 1924. AASLD 2017. Hepatology; 66:1020A, 2017.
- [Result] Lau A, Joshi A, Nguyen AH, Gaggar A, Patterson SD, Woo J. Peripheral blood immune cell profiling in virally suppressed chronic hepatitis B (CHB) patients and CHB patients not on an oral antiviral therapy. HBV International Meeting 2017.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Asia, Europe, New Zealand, and North America. The first participant was screened on 10 November 2015. The last study visit occurred on 03 May 2019.
Pre-assignment Details: 260 participants were screened
Groups:
- TDF + Vesatolimod 1 mg: Main Study Phase: TDF 300 mg tablets orally once daily for up to 48 weeks + vesatolimod 1 mg tablet orally once a week (every 7 days) for 12 doses.
  Optional Treatment Extension Phase: At Week 48 participants had the option to continue TDF 300 mg tablets orally once daily up to Week 144.
Period: Main Study Phase
Arm/Group | TDF + Placebo | TDF + Vesatolimod 1 mg | TDF + Vesatolimod 2 mg | TDF + Vesatolimod 4 mg
Started | 28 | 53 | 56 | 55
Completed | 28 | 53 | 54 | 52
Not Completed | 0 | 0 | 2 | 3
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0
Not completed — Withdrew Consent | 0 | 0 | 0 | 2
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1
Period: Optional Treatment Extension Phase(OTEP)
Arm/Group | TDF + Placebo | TDF + Vesatolimod 1 mg | TDF + Vesatolimod 2 mg | TDF + Vesatolimod 4 mg
Started | 27 (1 participant who completed the Main Study Phase did not enter the OTEP.) | 51 (2 participants who completed the Main Study Phase did not enter the OTEP.) | 54 | 49 (3 participants who completed the Main Study Phase did not enter the OTEP.)
Completed | 26 | 44 | 50 | 44
Not Completed | 1 | 7 | 4 | 5
Not completed — Withdrew Consent | 0 | 3 | 1 | 4
Not completed — Investigator's discretion | 1 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Pregnancy | 0 | 1 | 0 | 0
Not completed — Non-compliance with Study Drug | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who took at least 1 dose of study drug.
Groups:
- TDF + Placebo: Main Study Phase: TDF 300 mg tablets orally once daily for up to 48 weeks + placebo administered orally once a week (every 7 days) for 12 doses.
  Optional Treatment Extension Phase: At Week 48 participants had the option to continue TDF 300 mg tablets orally once daily up to Week 144.
- Total: Total of all reporting groups
Arm/Group | TDF + Placebo | TDF + Vesatolimod 1 mg | TDF + Vesatolimod 2 mg | TDF + Vesatolimod 4 mg | Total
Number analyzed (Participants) | 28 | 53 | 56 | 55 | 192
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (10.4) | 41 (9.6) | 44 (10.3) | 44 (10.3) | 42 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 21 | 16 | 20 | 69
  Male | 16 | 32 | 40 | 35 | 123
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 22 | 41 | 48 | 44 | 155
  Race: White | 4 | 6 | 5 | 10 | 25
  Race: Black or African American | 1 | 5 | 3 | 0 | 9
  Race: Native Hawaiian or Pacific Islander | 1 | 0 | 0 | 1 | 2
  Race: Other | 0 | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted = local regulators did not allow collection of race or ethnicity information.
  Participants
    Ethnicity: Hispanic or Latino | 0 | 0 | 0 | 0 | 0
    Ethnicity: Not Hispanic or Latino | 28 | 53 | 56 | 55 | 192
    Ethnicity: Not Permitted | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  New Zealand | 1 | 0 | 1 | 3 | 5
  Canada | 2 | 8 | 9 | 4 | 23
  South Korea | 7 | 12 | 17 | 15 | 51
  Hong Kong | 0 | 3 | 0 | 2 | 5
  United States | 6 | 14 | 13 | 10 | 43
  Taiwan | 5 | 4 | 6 | 6 | 21
  Italy | 6 | 8 | 6 | 12 | 32
  United Kingdom | 1 | 4 | 4 | 3 | 12
Serum Hepatitis B Surface Antigen (HBsAg) (log10 IU/mL) [Mean (Standard Deviation); unit: log10 IU/mL] | 3.8 (0.84) | 3.7 (0.84) | 3.5 (0.88) | 3.6 (0.74) | 3.6 (0.82)
Hepatitis B Envelope Antigen (HBeAg) Status [Count of Participants; unit: Participants]
  HBeAg Status- Negative | 17 | 33 | 33 | 34 | 117
  HBeAg Status- Positive | 11 | 20 | 23 | 21 | 75
Hepatitis B Virus (HBV) DNA [Mean (Standard Deviation); unit: log10 IU/mL] | 5.9 (2.10) | 5.9 (1.80) | 5.6 (1.85) | 5.9 (1.70) | 5.8 (1.82)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change (Measured in log10 IU/mL) in Hepatitis B Surface Antigen (HBsAg) From Baseline at Week 24
Description: The change from baseline to Week 24 in HBsAg (log10 IU/mL) was analyzed using a mixed model for repeated measures (MMRM). The model included treatment, baseline HBsAg (log10 IU/mL), baseline Hepatitis B Envelope Antigen (HBeAg) status (positive or negative), baseline alanine aminotransferase (ALT) level relative to upper limit of normal (ULN) (> 19 vs ≤ 19 IU/L for females; > 30 vs ≤ 30 IU/L for males), visit and treatment-by-visit interaction as fixed effects, and visit as a repeated measure.
Time Frame: Baseline; Week 24
Population: The Full Analysis Set included all participants who were randomized and took at least 1 dose of study drug.
Measure: Least Squares Mean (95% Confidence Interval); unit: log10 IU/mL
Groups:
- TDF + Placebo: Main Study Phase: TDF 300 mg tablets orally once daily for up to 48 weeks + Placebo administered orally once a week (every 7 days) for 12 doses.
- TDF + Vesatolimod 1 mg: Main Study Phase: TDF 300 mg tablets orally once daily for up to 48 weeks + vesatolimod 1 mg tablet orally once a week (every 7 days) for 12 doses.
- TDF + Vesatolimod 2 mg: Main Study Phase: TDF 300 mg tablets orally once daily for up to 48 weeks + vesatolimod 2 mg tablet orally once a week (every 7 days) for 12 doses.
- TDF + Vesatolimod 4 mg: Main Study Phase: TDF 300 mg tablets orally once daily for up to 48 weeks + vesatolimod 4 mg tablet orally once a week (every 7 days) for 12 doses.
Arm/Group | TDF + Placebo | TDF + Vesatolimod 1 mg | TDF + Vesatolimod 2 mg | TDF + Vesatolimod 4 mg
Number analyzed (Participants) | 28 | 53 | 54 | 54
log10 IU/mL | -0.163 [-0.305 to -0.022] | -0.056 [-0.159 to 0.047] | -0.146 [-0.246 to -0.045] | -0.036 [-0.138 to 0.065]
Statistical Analysis 1: Comparison: TDF + Placebo vs TDF + Vesatolimod 1 mg; Test type: Superiority; p = 0.227, MMRM — MMRM model included treatment, baseline ALT level, HBeAg baseline status, baseline HBsAg, visit and treatment-by-visit interaction as fixed effect and visit as repeated measurement; Least Squares Mean Difference = 0.107, 95% CI 2-sided [-0.067 to 0.282]
Statistical Analysis 2: Comparison: TDF + Placebo vs TDF + Vesatolimod 2 mg; Test type: Superiority; p = 0.840, MMRM — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.018, 95% CI 2-sided [-0.156 to 0.191]
Statistical Analysis 3: Comparison: TDF + Placebo vs TDF + Vesatolimod 4 mg; Test type: Superiority; p = 0.151, MMRM — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.127, 95% CI 2-sided [-0.047 to 0.301]

2. Secondary Outcome: Percentage of Participants With HBeAg Loss and Seroconversion at Week 24
Description: HBeAg loss was defined as qualitative HBeAg result changing from positive at baseline to negative at any postbaseline visit. HBeAg seroconversion was defined as qualitative Hepatitis B Envelope Antibody (HBeAb) result changing from negative at baseline to positive at any postbaseline visit. The Missing (M) = Failure (F) approach was used for this analysis.
Time Frame: Week 24
Population: Participants in the Full Analysis Set who were HBeAg positive at baseline were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | TDF + Placebo | TDF + Vesatolimod 1 mg | TDF + Vesatolimod 2 mg | TDF + Vesatolimod 4 mg
Number analyzed (Participants) | 11 | 20 | 23 | 21
percentage of participants | 0 | 0 | 0 | 0

3. Secondary Outcome: Percentage of Participants With HBeAg Loss and Seroconversion at Week 48
Description: HBeAg loss was defined as qualitative HBeAg result changing from positive at baseline to negative at any postbaseline visit. HBeAg seroconversion was defined as qualitative HBeAb result changing from negative at baseline to positive at any postbaseline visit. The Missing (M) = Failure (F) approach was used for this analysis.
Time Frame: Week 48
Population: Participants in the Full Analysis Set who were HBeAg positive at baseline were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | TDF + Placebo | TDF + Vesatolimod 1 mg | TDF + Vesatolimod 2 mg | TDF + Vesatolimod 4 mg
Number analyzed (Participants) | 11 | 20 | 23 | 21
percentage of participants | 0 | 5.0 | 4.3 | 4.8

4. Secondary Outcome: Percentage of Participants With HBsAg Loss and Seroconversion at Week 24
Description: HBsAg loss was defined as qualitative HBsAg result changing from positive at baseline to negative at any postbaseline visit. HBsAg seroconversion was defined as qualitative Hepatitis B Surface Antibody (HBsAb) result changing from negative at baseline to positive at any postbaseline visit. The Missing (M) = Failure (F) approach was used for this analysis.
Time Frame: Week 24
Population: Participants in the Full Analysis Set who were HBsAg positive at baseline were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | TDF + Placebo | TDF + Vesatolimod 1 mg | TDF + Vesatolimod 2 mg | TDF + Vesatolimod 4 mg
Number analyzed (Participants) | 28 | 53 | 56 | 55
percentage of participants | 0 | 0 | 0 | 0

5. Secondary Outcome: Percentage of Participants With HBsAg Loss and Seroconversion at Week 48
Description: HBsAg loss was defined as qualitative HBsAg result changing from positive at baseline to negative at any postbaseline visit. HBsAg seroconversion was defined as qualitative HBsAb result changing from negative at baseline to positive at any postbaseline visit. The Missing (M) = Failure (F) approach was used for this analysis.
Time Frame: Week 48
Population: Participants in the Full Analysis Set who were HBsAg positive at baseline were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | TDF + Placebo | TDF + Vesatolimod 1 mg | TDF + Vesatolimod 2 mg | TDF + Vesatolimod 4 mg
Number analyzed (Participants) | 28 | 53 | 56 | 55
percentage of participants | 0 | 0 | 0 | 0

6. Secondary Outcome: Mean Change (Measured in log10 IU/mL) in HBsAg From Baseline at Week 12
Time Frame: Baseline; Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | TDF + Placebo | TDF + Vesatolimod 1 mg | TDF + Vesatolimod 2 mg | TDF + Vesatolimod 4 mg
Number analyzed (Participants) | 27 | 53 | 55 | 52
log10 IU/mL | -0.087 (0.2199) | -0.041 (0.2283) | -0.138 (0.5247) | -0.020 (0.2668)

7. Secondary Outcome: Mean Change (Measured in log10 IU/mL) in HBsAg From Baseline at Week 48
Time Frame: Baseline; Week 48
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | TDF + Placebo | TDF + Vesatolimod 1 mg | TDF + Vesatolimod 2 mg | TDF + Vesatolimod 4 mg
Number analyzed (Participants) | 28 | 53 | 54 | 53
log10 IU/mL | -0.338 (0.8922) | -0.079 (0.2912) | -0.197 (0.5757) | -0.088 (0.3700)

8. Secondary Outcome: Percentage of Participants With a ≥ 0.5 log10 IU/mL Decline in Serum HBsAg Titers From Baseline at Week 12
Description: HBsAg ≥ 0.5 log10 IU/mL decline was defined as a decline from baseline in log10 IU/mL serum HBsAg ≥ 0.5 at the Week 12 post-baseline visit. Missing values were considered failures.
Time Frame: Baseline to Week 12
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | TDF + Placebo | TDF + Vesatolimod 1 mg | TDF + Vesatolimod 2 mg | TDF + Vesatolimod 4 mg
Number analyzed (Participants) | 28 | 53 | 56 | 55
percentage of participants | 7.1 | 3.8 | 10.7 | 1.8

9. Secondary Outcome: Percentage of Participants With a ≥ 0.5 log10 IU/mL Decline in Serum HBsAg Titers From Baseline at Week 24
Description: HBsAg ≥ 0.5 log10 IU/mL decline was defined as a decline from baseline in log10 IU/mL serum HBsAg ≥ 0.5 at the Week 24 post-baseline visit.
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | TDF + Placebo | TDF + Vesatolimod 1 mg | TDF + Vesatolimod 2 mg | TDF + Vesatolimod 4 mg
Number analyzed (Participants) | 28 | 53 | 56 | 55
percentage of participants | 10.7 | 3.8 | 10.7 | 3.6

10. Secondary Outcome: Percentage of Participants With a ≥ 0.5 log10 IU/mL Decline in Serum HBsAg Titers From Baseline at Week 48
Description: as for outcome 8
Time Frame: Baseline to Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | TDF + Placebo | TDF + Vesatolimod 1 mg | TDF + Vesatolimod 2 mg | TDF + Vesatolimod 4 mg
Number analyzed (Participants) | 28 | 53 | 56 | 55
percentage of participants | 17.9 | 5.7 | 16.1 | 14.5

11. Secondary Outcome: Percentage of Participants With Hepatitis B Virus Deoxyribonucleic Acid (HBV DNA) < Lower Limit of Quantitation (LLOQ) at Week 24
Description: LLOQ for HBV DNA was defined as 20 IU/mL. The participants with missing information were excluded from the analysis.
Time Frame: Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | TDF + Placebo | TDF + Vesatolimod 1 mg | TDF + Vesatolimod 2 mg | TDF + Vesatolimod 4 mg
Number analyzed (Participants) | 28 | 53 | 56 | 55
percentage of participants | 53.6 | 58.5 | 59.3 | 63.0

12. Secondary Outcome: Percentage of Participants With HBV DNA < LLOQ at Week 48
Description: LLOQ for HBV DNA was defined as 20 IU/mL. The participants with missing information were excluded from the analysis.
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | TDF + Placebo | TDF + Vesatolimod 1 mg | TDF + Vesatolimod 2 mg | TDF + Vesatolimod 4 mg
Number analyzed (Participants) | 28 | 53 | 56 | 55
percentage of participants | 64.3 | 62.3 | 75.9 | 75.5

13. Secondary Outcome: Percentage of Participants Experiencing Virologic Breakthrough
Description: Virologic breakthrough was defined as confirmed HBV DNA ≥ 69 IU/mL after having had HBV DNA < 69 IU/mL or confirmed 1.0 log10 IU/mL or greater increase in HBV DNA from nadir. Confirmation requires 2 consecutive occurrences of elevation in HBV DNA to > 69 IU/mL after having had HBV DNA < 69 IU/mL or 1.0 log10 IU/mL or greater increases in HBV DNA from nadir.
Time Frame: Weeks 24 and 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | TDF + Placebo | TDF + Vesatolimod 1 mg | TDF + Vesatolimod 2 mg | TDF + Vesatolimod 4 mg
Number analyzed (Participants) | 28 | 53 | 56 | 55
percentage of participants
  Week 24 | 0 | 0 | 1.8 | 0
  Week 48 | 0 | 3.8 | 1.8 | 0

14. Secondary Outcome: Number of Participants With Sequence Changes From Baseline Within the HBV Polymerase/Reverse Transcriptase (Pol/RT)
Description: Sequence analysis of the HBV pol/RT was attempted for any participant who had HBV DNA ≥ 69 IU/mL at Week 48 or early discontinuation. Results of the alignment of Week 48 and baseline sequence were reported as a change from baseline sequence.
Time Frame: Baseline; Week 48
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | TDF + Placebo | TDF + Vesatolimod 1 mg | TDF + Vesatolimod 2 mg | TDF + Vesatolimod 4 mg
Number analyzed (Participants) | 5 | 13 | 5 | 7
Participants | 2 | 4 | 2 | 2

15. Secondary Outcome: Pharmacokinetic (PK) Parameter: AUClast of Vesatolimod
Description: AUClast is defined as the area under the concentration versus time curve from time zero to the last quantifiable concentration.
Time Frame: Week 11: Predose, 0.5, 1, 2, 4, 6, 8, 10, 12, and 24 hours postdose
Population: The PK Substudy Analysis Set included all randomized participants who took at least 1 dose of vesatolimod, participated in the PK substudy, and had at least 1 non-missing steady state PK parameter.
Measure: Mean (Standard Deviation); unit: hour*picogram/milliliter (h*pg/mL)
Arm/Group | TDF + Vesatolimod 1 mg | TDF + Vesatolimod 2 mg | TDF + Vesatolimod 4 mg
Number analyzed (Participants) | 5 | 5 | 4
hour*picogram/milliliter (h*pg/mL) | 5252.3 (5756.26) | 7170.6 (4569.83) | 28537.2 (23608.94)

16. Secondary Outcome: PK Parameter: AUCinf of Vesatolimod
Description: AUCinf is defined as the concentration of drug extrapolated to infinite time.
Time Frame: Week 11: Predose, 0.5, 1, 2, 4, 6, 8, 10, 12, and 24 hours postdose
Population: Participants in the PK Substudy Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | TDF + Vesatolimod 1 mg | TDF + Vesatolimod 2 mg | TDF + Vesatolimod 4 mg
Number analyzed (Participants) | 5 | 5 | 4
h*pg/mL | 7277.3 (6550.71) | 10239.0 (6243.75) | 34534.8 (26482.89)

17. Secondary Outcome: PK Parameter: %AUCexp of Vesatolimod
Description: %AUCexp is defined as the percentage of AUC extrapolated between AUClast and AUCinf.
Time Frame: Week 11: Predose, 0.5, 1, 2, 4, 6, 8, 10, 12, and 24 hours postdose
Population: Participants in the PK Substudy Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of AUC
Arm/Group | TDF + Vesatolimod 1 mg | TDF + Vesatolimod 2 mg | TDF + Vesatolimod 4 mg
Number analyzed (Participants) | 5 | 5 | 4
Percentage of AUC | 31.1 (19.70) | 28.6 (11.42) | 19.3 (6.15)

18. Secondary Outcome: PK Parameter: Cmax of Vesatolimod
Description: Cmax is defined as the maximum concentration of drug.
Time Frame: Week 11: Predose, 0.5, 1, 2, 4, 6, 8, 10, 12, and 24 hours postdose
Population: Participants in the PK Substudy Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: picogram/milliliter (pg/mL)
Arm/Group | TDF + Vesatolimod 1 mg | TDF + Vesatolimod 2 mg | TDF + Vesatolimod 4 mg
Number analyzed (Participants) | 5 | 5 | 4
picogram/milliliter (pg/mL) | 667.8 (785.44) | 850.4 (569.75) | 4957.5 (5035.46)

19. Secondary Outcome: PK Parameter: Clast of Vesatolimod
Description: Clast is defined as the last observable concentration of drug.
Time Frame: Week 11: Predose, 0.5, 1, 2, 4, 6, 8, 10, 12, and 24 hours postdose
Population: Participants in the PK Substudy Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | TDF + Vesatolimod 1 mg | TDF + Vesatolimod 2 mg | TDF + Vesatolimod 4 mg
Number analyzed (Participants) | 5 | 5 | 4
pg/mL | 92.8 (73.80) | 119.0 (74.45) | 328.0 (165.19)

20. Secondary Outcome: PK Parameter: Tmax of Vesatolimod
Description: Tmax is defined as the time (observed time point) of Cmax
Time Frame: Week 11: Predose, 0.5, 1, 2, 4, 6, 8, 10, 12, and 24 hours postdose
Population: Participants in the PK Substudy Analysis Set were analyzed.
Measure: Median (Full Range); unit: hours
Arm/Group | TDF + Vesatolimod 1 mg | TDF + Vesatolimod 2 mg | TDF + Vesatolimod 4 mg
Number analyzed (Participants) | 5 | 5 | 4
hours | 1.00 [0.47 to 4.00] | 2.00 [2.00 to 4.00] | 3.00 [1.00 to 4.00]

21. Secondary Outcome: PK Parameter: Tlast of Vesatolimod
Description: Tlast is defined as the time (observed time point) of Clast.
Time Frame: Week 11: Predose, 0.5, 1, 2, 4, 6, 8, 10, 12, and 24 hours postdose
Population: Participants in the PK Substudy Analysis Set were analyzed.
Measure: Median (Full Range); unit: hours
Arm/Group | TDF + Vesatolimod 1 mg | TDF + Vesatolimod 2 mg | TDF + Vesatolimod 4 mg
Number analyzed (Participants) | 5 | 5 | 4
hours | 24.00 [8.00 to 24.00] | 24.00 [24.00 to 24.00] | 24.00 [24.00 to 24.00]

22. Secondary Outcome: PK Parameter: T1/2 of Vesatolimod
Description: T1/2 is defined as the estimate of the terminal elimination half-life of the drug.
Time Frame: Week 11: Predose, 0.5, 1, 2, 4, 6, 8, 10, 12, and 24 hours postdose
Population: Participants in the PK Substudy Analysis Set were analyzed.
Measure: Median (Full Range); unit: hours
Arm/Group | TDF + Vesatolimod 1 mg | TDF + Vesatolimod 2 mg | TDF + Vesatolimod 4 mg
Number analyzed (Participants) | 5 | 5 | 4
hours | 10.79 [4.57 to 50.08] | 14.12 [12.32 to 26.49] | 13.32 [8.90 to 14.83]

23. Secondary Outcome: PK Parameter: CL/F of Vesatolimod
Description: CL/F is defined as the apparent oral clearance following administration of the drug.
Time Frame: Week 11: Predose, 0.5, 1, 2, 4, 6, 8, 10, 12, and 24 hours postdose
Population: Participants in the PK Substudy Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: liter/hour
Arm/Group | TDF + Vesatolimod 1 mg | TDF + Vesatolimod 2 mg | TDF + Vesatolimod 4 mg
Number analyzed (Participants) | 5 | 5 | 4
liter/hour | 273.9 (270.58) | 262.3 (144.45) | 156.2 (72.48)

ADVERSE EVENTS:
Time Frame: First dose date up to last dose of study drug (Maximum: 144 weeks)
Description: The Safety Analysis Set included all participants who took at least 1 dose of study drug.
Groups:
- TDF + Placebo: Main Study Phase: Tenofovir disoproxil fumarate (TDF) 300 mg tablets orally once daily for up to 48 weeks + placebo administered orally once a week (every 7 days) for 12 doses.
- TDF + Vesatolimod 1 mg: Main Study Phase: TDF 300 mg tablets orally once daily for up to 48 weeks + vesatolimod (GS 9620) 1 mg tablet orally once a week (every 7 days) for 12 doses.
- TDF Extension From TDF + Placebo: Optional Treatment Extension Phase: At Week 48 participants had the option to continue TDF 300 mg tablets orally once daily up to Week 144; Includes participants who received TDF + Placebo in the Main Study Phase.
- TDF Extension From TDF + Vesatolimod 1 mg: Optional Treatment Extension Phase: At Week 48 participants had the option to continue TDF 300 mg tablets orally once daily up to Week 144; includes participants who received TDF + Vesatolimod 1 mg in the Main Study Phase.
- TDF Extension From TDF + Vesatolimod 2 mg: Optional Treatment Extension Phase: At Week 48 participants had the option to continue TDF 300 mg tablets orally once daily up to Week 144; includes participants who received TDF + Vesatolimod 2 mg in the Main Study Phase.
- TDF Extension From TDF + Vesatolimod 4 mg: Optional Treatment Extension Phase: At Week 48 participants had the option to continue TDF 300 mg tablets orally once daily up to Week 144; includes participants who received TDF + Vesatolimod 4 mg in the Main Study Phase.
Arm/Group | TDF + Placebo | TDF + Vesatolimod 1 mg | TDF + Vesatolimod 2 mg | TDF + Vesatolimod 4 mg | TDF Extension From TDF + Placebo | TDF Extension From TDF + Vesatolimod 1 mg | TDF Extension From TDF + Vesatolimod 2 mg | TDF Extension From TDF + Vesatolimod 4 mg
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/53 | 0/56 | 0/55 | 0/27 | 0/51 | 0/54 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/28 | 1/53 | 1/56 | 1/55 | 1/27 | 4/51 | 5/54 | 1/49
Other Adverse Events (participants affected / at risk) | 14/28 | 25/53 | 27/56 | 33/55 | 7/27 | 14/51 | 13/54 | 12/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TDF + Placebo (N=28) | TDF + Vesatolimod 1 mg (N=53) | TDF + Vesatolimod 2 mg (N=56) | TDF + Vesatolimod 4 mg (N=55) | TDF Extension From TDF + Placebo (N=27) | TDF Extension From TDF + Vesatolimod 1 mg (N=51) | TDF Extension From TDF + Vesatolimod 2 mg (N=54) | TDF Extension From TDF + Vesatolimod 4 mg (N=49)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Adenomyosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pelvic congestion (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TDF + Placebo (N=28) | TDF + Vesatolimod 1 mg (N=53) | TDF + Vesatolimod 2 mg (N=56) | TDF + Vesatolimod 4 mg (N=55) | TDF Extension From TDF + Placebo (N=27) | TDF Extension From TDF + Vesatolimod 1 mg (N=51) | TDF Extension From TDF + Vesatolimod 2 mg (N=54) | TDF Extension From TDF + Vesatolimod 4 mg (N=49)
Abdominal distension (Gastrointestinal disorders) | 2 | 3 | 1 | 1 | 0 | 0 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 3 | 1 | 0 | 0 | 2 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 4 | 2 | 5 | 0 | 1 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 1 | 3 | 1 | 1 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 3 | 5 | 3 | 5 | 0 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 5 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 2 | 1 | 2 | 3 | 0 | 1 | 0 | 0
Chills (General disorders) | 1 | 2 | 6 | 10 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 6 | 8 | 6 | 14 | 0 | 2 | 1 | 2
Influenza like illness (General disorders) | 1 | 1 | 0 | 5 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 4 | 5 | 11 | 0 | 2 | 0 | 0
Gingivitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 2 | 2 | 1 | 0 | 5 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 3 | 0 | 4 | 2 | 3 | 4 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 3 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3 | 10 | 0 | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 4 | 2 | 2 | 2 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 5 | 4 | 9 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 3 | 1 | 5 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 5 | 4 | 10 | 12 | 0 | 2 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 2 | 2 | 2 | 1 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 1 | 1 | 1 | 0 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3 | 1 | 2 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years